CLINICAL TRIAL: NCT03406104
Title: Long-term Follow-up of ND4 LHON Subjects Treated With GS010 Ocular Gene Therapy in the RESCUE or REVERSE Phase III Clinical Trials (RESTORE)
Brief Title: RESCUE and REVERSE Long-term Follow-up
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-LHON-CLIN-06; 2017-002153-11 (EudraCT Number); NCT02652767 RESCUE (Other: clin.trial.gov); NCT02652780 REVERSE (Other: clin.trial.gov)
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Leber Hereditary Optic Neuropathy
Keywords: Heredity Optic Atrophy; Leber Hereditary Optic Atrophy; Leber Hereditary Optic Neuropathy; LHON; Eye Diseases; Hereditary Eye Diseases; Inborn Genetic Disease; Gene Therapy; Intravitreal Injections; Mitochondrial Disease; AAV2 Vectors; Nervous System Diseases; Neurodegenerative Disease; Heredodegenerative Disorders of the Nervous System
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Eye Diseases; Eye Diseases, Hereditary; Genetic Diseases, Inborn; Mitochondrial Diseases; Nervous System Diseases; Neurodegenerative Diseases | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: intra patient comparaison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GS010-treated Eyes (Experimental): Lenadogene nolparvovec Intravitreal ocular unilateral Injection Each participant will have one eye randomly selected to receive a single injection of GS010 and the other eye will receive a sham injection. GS010-treated Eyes: GS010 is a recombinant adeno-associated viral vector serotype 2 (rAAV2/2) containing the wild-type ND4 gene (rAAV2/2-ND4). Participants will receive a single dose of GS010 in one of their randomly selected eyes, via intravitreal injection containing 9E10 viral genomes in 90μL balanced salt solution (BSS) plus 0.001% Pluronic F68®.
  Interventions: Genetic: GS010
- Sham-treated Eyes (Sham Comparator): Sham Intravitreal ocular unilateral Injection Each participant will have one eye randomly selected to receive GS010 and the other eye will receive a sham injection. Eyes receiving sham injection will undergo the same preparatory procedures as eyes receiving GS010 injection, including pupillary dilation, topical anti-infection and topical anesthetic procedures. Sham intravitreal injection will be performed by applying pressure to the eye at the location of a typical intravitreal injection procedure using the blunt end of a syringe without a needle.
  Interventions: Other: Sham Intravitreal Injection

INTERVENTIONS:
Genetic: GS010 — Lenadogene nolparvovec Intravitreal ocular unilateral Injection
  Other Names: Lenadogene Nolparvovec
  Arms: GS010-treated Eyes
Other: Sham Intravitreal Injection — Lenadogene nolparvovec Intravitreal ocular unilateral Injection
  Arms: Sham-treated Eyes

SUMMARY:
The goal of this clinical trial is to assess the long-term safety and efficacy of GS010, a gene therapy, and assess the quality of life in subjects with LHON due to the G11778A ND4 mitochondrial mutation and who were treated in the Rescue or Reverse studies.

DETAILED DESCRIPTION:
Seven investigational centers from the RESCUE and REVERSE studies also participated in the RESTORE study, located in the European union and in the USA.

Primary objectives: to assess the long term safety of intravitreal injection up to 5 years of post treatment in subjects who were treated in the RESCUE or REVERSE studies.

Secondary objectives: (1) to assess the long-term efficacy of intravitreal GS010 administration up to 5 years post-treatment in subjects who were treated in the RESCUE or REVERSE studies; and (2) to assess the quality of life (QoL) in subjects who were treated with GS010 in the RESCUE or REVERSE studies for up to 5 years post-treatment.

Methodology: This was a Phase III prospective long-term follow-up (LTFU) clinical study of subjects previously treated with GS010 and Sham during 2 Phase III studies-RESCUE and REVERSE. The LTFU study followed subjects for an additional 3 years, for a total of 5 years post-injection. The LTFU study included 5 visits at 2, 2.5, 3, 4, and 5 years after the investigational medicinal product (IMP) injection. Safety, efficacy, and QoL variables were assessed during each of the 5 LTFU visits, and descriptive summaries and statistical testing were used for the analysis of the data.

This report presents the final analysis of results at Year 5 after treatment administration in RESCUE and REVERSE.

Number of analysed subjects: all subjects completing RECUE and REVERSE studies who provided consent for the RESTORE study: 62 subjects.

ELIGIBILITY:
Inclusion Criteria

* Subject was treated with GS010 IVT injection in either of the RESCUE or REVERSE Phase III clinical studies
* Subject of legal consent age has provided informed consent; subjects that are not of legal consent age have undergone their country-approved clinical trial enrollment consent process

Exclusion Criteria

* Subject is unwilling or unable to comply with the protocol requirements
* Subject has any medical or psychological condition that, in the opinion of the Investigator, may compromise his or her safe participation in the study
* Subject is taking or intending to take idebenone during the long-term follow-up study period

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Newman, MD, Principal Investigator — Emory University Hospital Atlanta, Georgia, United States, 30322
Locations (7):
- United States (3):
  - Doheny Eye Center UCLA, Pasadena, California
  - Emory University Hospital, Atlanta, Georgia
  - Wills Eye Institute, Philadelphia, Pennsylvania
- CHNO Les Quinze Vingts, Paris, France
- LMU Klinikum der Universität München / Friedrich-Baur-Institut, Munich, Germany
- Ospedale Bellaria, Bologna, Italy
- Moorfields Eye Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Yu-Wai-Man P, Newman NJ, Biousse V, Carelli V, Moster ML, Vignal-Clermont C, Klopstock T, Sadun AA, Sergott RC, Hage R, Degli Esposti S, La Morgia C, Priglinger C, Karanja R, Taiel M, Sahel JA; LHON Study Group. Five-Year Outcomes of Lenadogene Nolparvovec Gene Therapy in Leber Hereditary Optic Neuropathy. JAMA Ophthalmol. 2025 Feb 1;143(2):99-108. doi: 10.1001/jamaophthalmol.2024.5375. PMID 39699886
- [Derived] Carelli V, Newman NJ, Yu-Wai-Man P, Biousse V, Moster ML, Subramanian PS, Vignal-Clermont C, Wang AG, Donahue SP, Leroy BP, Sergott RC, Klopstock T, Sadun AA, Rebolleda Fernandez G, Chwalisz BK, Banik R, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA; the LHON Study Group. Indirect Comparison of Lenadogene Nolparvovec Gene Therapy Versus Natural History in Patients with Leber Hereditary Optic Neuropathy Carrying the m.11778G>A MT-ND4 Mutation. Ophthalmol Ther. 2023 Feb;12(1):401-429. doi: 10.1007/s40123-022-00611-x. Epub 2022 Nov 30. PMID 36449262
- [Derived] Newman NJ, Yu-Wai-Man P, Carelli V, Biousse V, Moster ML, Vignal-Clermont C, Sergott RC, Klopstock T, Sadun AA, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA. Intravitreal Gene Therapy vs. Natural History in Patients With Leber Hereditary Optic Neuropathy Carrying the m.11778G>A ND4 Mutation: Systematic Review and Indirect Comparison. Front Neurol. 2021 May 24;12:662838. doi: 10.3389/fneur.2021.662838. eCollection 2021. PMID 34108929

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patient Treated in RECUE and REVERSE Studies: all patients previously treated in RESCUE and REVERSE studies entered in this long term follow up study.
Period: Overall Study
Arm/Group | All Patient Treated in RECUE and REVERSE Studies
Started | 62
Completed | 55
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — due to Covid patient did not want to travel | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Groups:
- Lenadogene Nolparvovec and Sham All Participants: All participants who were enrolled and received both study treatments, GS010 and Sham. All participants in the study received both GS010 and the sham procedure simultaneously. Participants were randomly assigned to receive GS010 in either the right or left eye. The same participants also received the sham procedure in the eye not assigned to GS010, at the same study visit.
  GS010: Either the right or left eye received one single dose of GS010 (9E10 vg/eye) via an intravitreal (IVT) injection. The volume of the injected formula was 90 µL. The injection was performed in the vitreous humor under local anesthesia.
  Sham procedure: Either the right or left eye (the eye not randomly assigned to GS010) received the sham procedure. One single sham IVT injection was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
Arm/Group | Lenadogene Nolparvovec and Sham All Participants
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 55
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31
  Italy | 1
  United Kingdom | 5
  France | 16
  Germany | 9
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: LogMAR] — Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity scale.
  LogMAR | 1.40 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Adverse Events (AEs)
Description: Number of Eyes with Ocular Adverse events related to study treatment or study procedures as judged by the investigator reported from year 2 to year 5 post treatment
Time Frame: from year 2 to year 5 post treatment
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- GS010 Treated Eyes: All eyes that received the study treatment, GS010. Each participant was randomly assigned GS010 in either the right or left eye. The eye assigned to GS010 received one single dose of GS010 (9E10 vg/eye) via an intravitreal (IVT) injection. The volume of the injected formula was 90 μL. The injection was performed in the vitreous humor under local anesthesia.
  The same participants also received the sham procedure in the right or left eye, which was not assigned to receive GS010, at the same study visit.
- Sham Treated Eyes: All eyes that received the Sham. Each participant was randomly assigned GS010 in either the right or left eye, the eye not assigned GS010 received the sham procedure. The eye assigned to the Sham received one single sham intravitreal (IVT) injection, which was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
  The same participants also received GS010 in the right or left eye, which did not receive the sham procedure, at the same study visit.
Arm/Group | GS010 Treated Eyes | Sham Treated Eyes
Number analyzed (Participants) | 62 | 62
Number analyzed (eyes) | 62 | 62
eyes | 5 | 1

2. Secondary Outcome: Visual Acuity
Description: Change from Nadir to 5 Years post-treatment, Assessed at Baseline in RESCUE and REVERSE studies to year 5 post-treatment, expressed in LogMAR.
  On chart visual acuity: Visual acuity inferior or equal to LogMAR +1.6 Off chart visual acuity: Visual acuity superior to LogMar +1.7
  Normal vision LogMar: 0 and less than 0
Time Frame: Nadir to 5 Years post-treatment, Assessed at Baseline in RESCUE and REVERSE studies to year 5 post-treatment
Population: All efficacy analyses were conducted on the modified intent-to-treat population and additionally in subset populations, as appropriate.The modified intent-to-treat (mITT) population consisted of all subjects who received the IMP in RESCUE or REVERSE Phase III studies, consented to be enrolled in this LTFU study, and provided visual acuity data at Visit 2 (Year 2.5).
Measure: Mean (Standard Deviation); unit: LogMar
Units Other Than Participants: eyes
Arm/Group | GS010 Treated Eyes | Sham Treated Eyes
Number analyzed (Participants) | 62 | 62
Number analyzed (eyes) | 62 | 62
LogMar | -0.44 (0.46) | -0.39 (0.36)

3. Secondary Outcome: Responder Analysis: Clinically Relevant Recovery
Description: CRR clinically relevant recovery from Nadir defined as i/ for eyes on chart at Nadir, an improvement of at least -0.2 LogMar from Nadir and ii/ for eyes off chart at Nadir eyes that became on chart.
  Off chart visual acuity expressed in LogMar: more than +1.7 On chart visual acuity expressed in LogMar: less than 1.6 Normal vision LogMar: 0 and less than 0
Time Frame: Nadir to 5 Years post-treatment, Assessed at Baseline in RESCUE and REVERSE studies to year 5 post-treatment
Population: as for outcome 2
Measure: Number; unit: percentage of eye
Units Other Than Participants: eyes
Arm/Group | GS010 Treated Eyes | Sham Treated Eyes
Number analyzed (Participants) | 62 | 62
Number analyzed (eyes) | 62 | 62
percentage of eye | 60 | 66

4. Other Pre Specified Outcome: Eyes on Chart
Description: Definition: Visual acuity inferior or equal to LogMAR +1.6 at 5 Years post treatment
Time Frame: Year 5 post-treatment
Population: as for outcome 2
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 62 | 62
Number analyzed (eyes) | 62 | 62
percentage of eyes | 76 | 79

ADVERSE EVENTS:
Time Frame: from 2 to 5 years
Groups:
- Subjects: All eyes that received the Sham. Each participant was randomly assigned GS010 in either the right or left eye, the eye not assigned GS010 received the sham procedure. The eye assigned to the Sham received one single sham intravitreal (IVT) injection, which was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
  The same participants also received GS010 in the right or left eye, which did not receive the sham procedure, at the same study visit.
Arm/Group | Subjects
All-Cause Mortality (participants affected / at risk) | 2/62
Serious Adverse Events (participants affected / at risk) | 8/62
Other Adverse Events (participants affected / at risk) | 19/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects (N=62)
hip fracture (Injury, poisoning and procedural complications) | 2 (2)
humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1)
lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
limb injury (Injury, poisoning and procedural complications) | 1 (1)
cerebral haemorrage (Nervous system disorders) | 1 (1)
glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
appenditis perforated (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects (N=62)
Cataract (Eye disorders) | 6 (13)
Gamma-Glutamyltransferase Increased (Investigations) | 5 (5)
Intraocular Pressure Increased (Eye disorders) | 4 (8)
Covid-19 (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03406104/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03406104/SAP_001.pdf